CLINICAL TRIAL: NCT01012466
Title: The Physical Effects of Pain Catastrophizing on Normal Labor
Brief Title: The Physical Effects of Pain Catastrophizing in Labor
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Beth Darnall, PhD, Principal Investigator, Oregon Health and Science University
Other Study IDs: 5203; 5K12HD04348807
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy
Keywords: pregnancy; birth; labor; labor pain; catastrophizing
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether labor self-efficacy (as determined by scores for the Lederman PSEQ II (self-efficacy scores) impacts the second stage 2 length (nromal vs. prolonged) as determined by quartile ranges for our sample. Other studies have shown that women who experience intense pain in the earliest stages of labor have a higher risk of complications. The investigators want to know if negative thoughts can predict this outcome.

DETAILED DESCRIPTION:
Subjects will complete questionnaires at three timepoints: during the prenatal period, within 24-48 hours of giving birth, and 4-8 weeks postpartum. The questionnaires will measure pain catastrophizing, depression, maternal support, support and control in birth, and childbirth satisfaction. Chart review following delivery will record data such as length of labor, medication used, need for augmentation or surgical delivery, complications.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 weeks of pregnancy
* Nulliparous
* Singleton pregnancy
* Low risk pregnancy

Exclusion Criteria:

* Primiparous and multiparous women
* Women who request cesarean delivery
* Women who are pregnant with twins
* Women who plan induction
* Women who deliver before 37 weeks
* Women enrolled in the "Centering Pregnancy" program at the Family Birth Center
* High risk pregnancies
* Severe mental illness that impairs cognition or function
* Suicidal ideation
* Women who do not speak English or Spanish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nulliparous women attending the prenatal clinic at Oregon Health & Science University
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Relationship between pain catastrophizing and abnormal labor (deviation of progress in labor from norms) | Immediate postpartum

SECONDARY OUTCOMES:
Relationship between pain catastrophizing and reported pain in labor | 1 day postpartum and 4-8 weeks postpartum
Relationship between pain catastrophizing and satisfaction with birth experience and care | 1 day postpartum and 4-8 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States